CLINICAL TRIAL: NCT02741648
Title: Red Blood Cell Transfusion and Digestive Tract Oxygenation in Preterm Infants Weighing ≤ 1250 Grams
Brief Title: RBC Irradiation, Anemia and Gut Injury
Acronym: RBC-mNIRS
Status: Active, not recruiting | Type: Observational
Sponsor: Emory University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Ravi Mangal Patel, Professor, Emory University
Other Study IDs: IRB00083691; 2P01HL086773 (NIH); 1R01HL138714 (NIH); 2025P010798 (Other: Emory IRB)
Record Dates: First submitted 2016-04-13; First posted 2016-04-18 (Estimated); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Anemia; Necrotizing Enterocolitis
Keywords: Red Blood Cell Transfusion; Digestive tract problems; Extremely Low Birth Weight
MeSH Terms: conditions — Anemia; Enterocolitis, Necrotizing | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Residual patient blood samples (obtained for routine clinical testing), urine, stool and breast milk will be collected, frozen and stored. If a baby develops a digestive tract complication, the stored specimens will be studied in the laboratory in an effort to identify markers of a healthy digestive tract versus illness.
  A sample of transfused RBCs will be obtained from the RBC unit at each RBC transfusion. If the baby develops a digestive tract complication the stored specimens will be studied in the laboratory to identify changes in the biochemical compounds of the transfused blood that may have taken place over time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (4):
- ELBW Infants with Prolonged Irradiation Storage Time: Extremely Low Birth Weight Infants whose Red Blood Cell (RBC) transfusion had prolonged Irradiation Storage Time (IST) being tested with metabolomics profile.
  Interventions: Device: Near Infrared Spectroscopy
- ELBW Infants without Irradiation Storage: Extremely Low Birth Weight Infants whose Red Blood Cell (RBC) transfusion did not have Irradiation Storage being tested with metabolomics profile.
  Interventions: Device: Near Infrared Spectroscopy
- ELBW Infants Reaching the NEC Window: Extremely low birth weight infants who reach 28 to 34 postmenstrual week age, which is the NEC window.
  Interventions: Other: Non-invasive Image-based Anemia Assessment
- ELBW Infants: Extremely low birth weight infants having intestinal microbial profiles examined via stool collected from discarded diapers, and immune cell function and serum cytokine levels examined using residual blood.

INTERVENTIONS:
Device: Near Infrared Spectroscopy — INVOS 5100C Cerebral/Somatic Oximeter is an FDA-approved device used to measure renal and mesenteric tissue oxygenation, as defined by regional oxygenation saturation levels (rSO2). Two probe site monitoring will be used to evaluate differential tissue bed oxygenation. Adhesive sensor probes are applied to the periumbilical area for mesenteric monitoring and to the flank area for renal monitoring.
  Other Names: NIRS
  Groups: ELBW Infants with Prolonged Irradiation Storage Time; ELBW Infants without Irradiation Storage
Other: Non-invasive Image-based Anemia Assessment — A trained research associate will take 2 images (one with the camera flash on and one with the camera flash off) of the patient's fingernail beds, toe nail beds, palm of the hand and sole of the foot. Images will be taken within 24 hours, preceding, or following, each complete blood count (CBC) collection on each consented patient. The anemia diagnosing algorithm will then be run on the images.
  Groups: ELBW Infants Reaching the NEC Window

SUMMARY:
The purpose of this trial is to study the effect that anemia and red blood cell (RBC) transfusions have on oxygen levels in the digestive tracts of extremely low birth weight (ELBW) infants and to look for possible markers in a baby's blood, urine and/or stool that may lead to a better understanding of what makes an ELBW infant at risk for digestive tract problems such as necrotizing enterocolitis.

DETAILED DESCRIPTION:
Necrotizing Enterocolitis (NEC) is a leading cause of neonatal morbidity and mortality in preterm infants. To date, no effective genetic or clinical markers exist to predict which premature infant will develop NEC, limiting targeted prevention strategies. Anemia and digestive tract complications are common problems in extremely low birth weight infants. Anemia is a condition in which the body does not have enough red blood cells (RBC). RBCs are important because they contain hemoglobin, the substance that carries oxygen throughout the body. Transfusions of RBCs in these infants is frequently required to correct the anemia.

Multiple observational studies have reported an association between the exposure to red blood cell (RBC) transfusion and the subsequent development of transfusion related-NEC (TR-NEC).However, no clinical studies have investigated the underlying pathophysiologic mechanisms of TR-NEC. In adults, prolonged RBC storage prior to transfusion has been associated with adverse outcomes and may also contribute to TR-NEC. However, the chronological storage age of blood may not be an accurate gauge of donor RBC function; irradiation of RBCs to prevent transfusion-associated graft-vs-host disease may also contribute to TR-NEC. Currently, the duration considered safe for RBC storage following irradiation (irradiation storage time (IST)) is unclear. Given the multifactorial etiology of NEC, preventative efforts will be more successful if clinicians understand the underlying pathophysiologic mechanisms and modifiable risk factors.

In this study the researchers will conduct a multicenter observational cohort study of very preterm (VPT) infants weighing ≤1250g at birth to prospectively investigate the associations between RBC transfusion, digestive tract oxygenation, and TR-NEC. The overarching hypothesis for this study is that irradiation of RBC units followed by prolonged storage perturbs RBC metabolism and function, and these derangements are associated with paradoxical microvascular vasoconstriction, tissue hypoxia and TR-NEC in transfused infants with already impaired gut oxygenation due to significant anemia. All RBC units transfused to VPT infants throughout the study will be stored based on current standard operating procedures per local site blood banking practices. There will be no study-specific approaches to transfusions or transfusion thresholds, and the decision to transfusion will be made as part of current clinical care by the treating clinicians. No study-specific blood draws will occur and all samples will be obtained from residual samples collected for clinical care that are to be discarded.

Oxygen levels in the digestive tract will be measured before, during and after each blood transfusion using a tissue oxygen monitor called Near Infrared Spectroscopy (NIRS). By using this technology, the researchers intend to better understand intestinal blood flow patterns. RBC function in RBC products transfused to infants will be compared between the infants who develop TR-NEC and matched control infants who do not develop TR-NEC. The researchers will explore the clinical implications of severe anemia when infants are 28 to 34 weeks of postmenstrual age, which is when infants are vulnerable to NEC.

Currently, there are no inexpensive, simple, patient/healthcare provider-operated hemoglobin tests available for diagnosing and assessing the degree of anemia without the use of a blood draw. To that end, Emory investigators have recently developed an algorithm that enables patients/healthcare providers to check if a patient is anemic by simply taking a picture of their fingernail beds on a Smartphone, and running the algorithm on a computer using MATLAB. These studies have shown that the degree of pallor in the fingernail beds, correlates with physiologic levels of hemoglobin in the blood and determines whether or not the patient is anemic. To date, the accuracy of this device has only been tested on adults and older children. Having an accurate and noninvasive means of testing for anemia in VPT infants would reduce the number of blood draws required, decrease the common side effects of phlebotomy, transfusion of RBCs, and would potentially be more cost-effective. As an additional study aim, the researchers of this study seek to develop a new image analysis algorithm (IAA) to predict hemoglobin level and anemia status from fingernail photos. The fingernail beds of VPT infants are extremely small and therefore it is uncertain if the nail bed is the most accurate site to assess anemia in these infants. To determine which site is most accurate in this population pictures will be taken of the fingernail beds, the toe nail beds, the palm of the hand and the sole of the foot with be photographed and analyzed.

Leftover samples of blood, urine, stool, and breast milk will be frozen, and stored and in the event a baby develops a digestive tract complication the samples will be studied in a laboratory to identify markers that indicate a healthy digestive tract versus illness. Immune cell function, digestive tract microbial changes, and serum cytokine levels will be compared between very preterm infants who develop NEC and those who do not.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight ≤1250 grams
* Postnatal age within 7 days of birth

Exclusion Criteria:

* Infant not expected to live beyond 7 days of life based on assessment of treating neonatologist
* Severe congenital abnormality expected to affect life expectancy
* RBC or platelet transfusion at an outside institution occurring prior to screening
* Maternal refusal to participate

Ages: 1 Day to 5 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Extremely low birth weight newborn infants born at Emory University Hospital Midtown, Grady Health System, and Northside Hospital Neonatology. Infants will be followed at Children's Healthcare of Atlanta.
Sampling Method: Non-Probability Sample
Enrollment: 324 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Mesenteric Tissue Oxygenation | 60 Minutes prior to transfusion to 48 hours after transfusion
  Mesenteric tissue oxygenation is measured in infants receiving RBC transfusion. Mesenteric regional saturation of oxygen (MES-rSO2) levels are measured via the INVOS 5100C Cerebral/Somatic Oximeter by applying an adhesive sensor probe to the patient's periumbilical area for mesenteric monitoring. MES-rSO2 will be compared between infants receiving RBC transfusion with and without IST.
Infants Developing TR-NEC | 60 Minutes prior to transfusion to 48 hours after transfusion
  Development of TR-NEC will be compared between infants receiving RBC transfusion with and without IST.
Inhibition of NO-Mediated Vasodilation | 60 Minutes prior to transfusion to 48 hours after transfusion
  Inhibition of NO-mediated vasodilation will be used to assess RBC function among transfused infants who develop TR-NEC and matched control infants who do not develop TR-NEC.
Metabolic Changes of Red Blood Cells | 60 Minutes prior to transfusion to 48 hours after transfusion
  Functional defects of transfused RBCs will be examined to assess metabolic changes of RBCs among transfused infants who develop TR-NEC and matched control infants who do not develop TR-NEC.
Mesenteric Tissue Oxygenation During the NEC Window Period | 28 to 34 Weeks Post Menstrual Age
  ELBW infants that reach the window when NEC typically occurs will be further compared as those with vs without anemia. Regional Oxygenation Saturation Levels (rSO2) are measured via the INVOS 5100C Cerebral/Somatic Oximeter by applying an adhesive sensor probe to the patient's periumbilical area for mesenteric monitoring. NIRS will be performed once per week (whether transfused or not) for a 48 hour period starting each Monday (day of routine lab draw to evaluate anemia).
Immune Cell Function | Up to 90 days of age
  Anemia significantly modulates immune function and may predispose infants to NEC through alterations in T cell activation and the presence of immunomodulatory erythroid precursors. Immune cell function profiles will be compared between infants who develop TR-NEC and matched controls who do not.
Microbial Changes | Up to 90 days of age
  Alterations in the microbiota may further drive dysregulated immune function toward increased overall inflammation and the development of NEC. Microbial profiles will be compared between infants who develop TR-NEC and matched controls who do not.
Serum Cytokine Levels | Up to 90 days of age
  Serum cytokine levels will be compared between infants who develop TR-NEC and matched controls who do not.

OTHER OUTCOMES:
Image Analysis Algorithm | Up to 90 days of age
  The researchers will use an image analysis algorithm (IAA) to examine structural information in fingernail photos and image metadata to accurately predict hemoglobin level and anemia status.
Development of a Clustering Method for Identification of Anemia | Up to 90 days of age
  The researchers will develop a new clustering method for further understanding sub-population structures of fingernail photos and image megadata to identify subgroups of infants with high anemia risk.
Image Analysis Algorithm | Up to 90 days of age
  The researchers will develop a new clustering method for further understanding sub-population structures of fingernail photos and image megadata to identify subgroups of infants with high anemia risk.

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Patel, MD, MSc, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Grady Memorial Hospital, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Northside Hospital - Neonatology, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marin T, Patel RM, Roback JD, Stowell SR, Guo Y, Easley K, Warnock M, Skvarich J, Josephson CD. Does red blood cell irradiation and/or anemia trigger intestinal injury in premature infants with birth weight </= 1250 g? An observational birth cohort study. BMC Pediatr. 2018 Aug 11;18(1):270. doi: 10.1186/s12887-018-1241-5. PMID 30098602